CLINICAL TRIAL: NCT00395005
Title: The Correlation of Urine Tissue Kallikrein Protein Level With Cytokines, Degree of Proteinuria and Renal Function Deterioration in Chronic Renal Disease Patients After Angiotensin II Receptor Blocking
Brief Title: Correlation of Urinary Kallikrein With Cytokines, Proteinuria and Renal Function in Chronic Renal Disease Patients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9561709146
Record Dates: First submitted 2006-10-31; First posted 2006-11-02 (Estimated); Last update posted 2007-03-23 (Estimated); Status verified 2006-10

CONDITIONS: Chronic Kidney Disease
Keywords: Kallikrein; Cytokines; Proteinuria; Renal function; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria

STUDY DESIGN:
Observational Model: Natural History | Time Perspective: Retrospective

SUMMARY:
Urinary kallikrein excretion is known to increase in patients with nephrotic syndrome and sick cell disease, but decrease in patients with chronic kidney disease or uremia. Some of authors consider urinary kallikrein is a marker of nephropathy. To evaluate the possible role of kallikrein kinin system in chronic kidney disease, we conduct a retrospective longitudinal observation study. Patients who participating in the "Efficacy of Pentoxifylline on Chronic Kidney Disease" study are included in the study. The morning spot urinary kallikrein and cytokines are measured at the time point of 0 and 12 month in addition to clinical parameters. The correlation of urinary kallikrein and cytokine concentration will be evaluated. Using multiple regression model, the relationship of urinary kallikrein excretion with degree of proteinuria, creatinine clearance and other clinical parameter will also be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* During June 2004 and June 2005 who participate the clinical study "Efficacy of Pentoxifylline on Chronic Kidney Disease" (ClinicalTrials.gov Identifier: NCT00155246)and sign the informed consent.
* Chronic kidney disease history > 3 months, Serum creatinine: 1.1~6.0 mg/dl in female. 1.3~6.2 mg/dl in male.
* Initial Random urine protein (mg/dl) /creatinine (mg/dl) ratio > 0.5

Exclusion Criteria:

* History of allergy to pentoxifylline;
* females are nursing or pregnant;
* Obstructive uropathy;
* Unable to stop chronic immunosuppressive therapy, NSAID;
* Congestive heart failure (New York Heart Association functional class III or IV);
* Unstable angina, myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention, within the past 6 months prior to signing the informed consent form;
* Cerebral hemorrhage within the past 6 months prior to signing the informed consent form;
* Retinal hemorrhage within the past 6 months prior to signing the informed consent form;
* Known or suspected secondary hypertension (e.g., primary aldosteronism, renovascular hypertension, pheochromocytoma);
* Severe uncontrolled hypertension with SBP > 220 mmHg and/or DBP > 115 mmHg;
* Hepatic dysfunction as defined by the following laboratory parameters: ALT or AST > 2 times the upper limit of the normal range;
* Biliary obstructive disorders (e.g. cholestasis);
* Active malignancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2006-10; Study Completion 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chih Chiang, MD, Principal Investigator — National Taiwan University Hospital